CLINICAL TRIAL: NCT02681458
Title: The Comparison of Dermatophytosis and Other Fungal Infections Between Drug Users and Non Drug Users
Brief Title: Superficial and Cutaneous Fungal Infections Among Drug-users in Northeast Region of Iran
Status: Completed | Type: Observational
Sponsor: Islamic Azad University of Mashhad (Other)
Responsible Party: Principal Investigator, Hassan Yazdanfar, Head of parasitology and mycology department, Islamic Azad University of Mashhad
Other Study IDs: IslamicAUM
Record Dates: First submitted 2016-01-31; First posted 2016-02-12 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Skin and Subcutaneous Tissue Fungal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — hair, nail, cutaneous lesions
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Drug Users: Case group that consisted of drug users with fungal infections
  Interventions: Other: Direct Examination
- Non-drug Users: Control group that consisted of non drug users with fungal infections
  Interventions: Other: Direct Examination

INTERVENTIONS:
Other: Direct Examination — It was an observational study and subjects received their routine treatment.

SUMMARY:
The purpose of this study was about survey of prevalence of fungal infections among drug users referring to methadone wards of Hospitals in northeast region of Iran

DETAILED DESCRIPTION:
There were two groups with overall members of 1436. Statistically, the investigators have used "Likelihood ratio " and " Exact's Fisher" tests.

ELIGIBILITY:
Inclusion Criteria:

* Suspected fungal lesions

Exclusion Criteria:

* non use of local or edible anti-fungal drugs and not taking bath within the last 48 hours of testing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: people from northeast region of Iran referring to Methadone clinics. there were no limitations of age and sex.
Sampling Method: Probability Sample
Enrollment: 1436 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Yazdanfar, MD, PhD, Study Chair — assistant professor of mycology and parasitology
Locations (1):
- Islamic Azad University of Mashhad, Mashhad, Khorasan Razavi, Iran

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided about this issue yet

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-drug Users: Control group that consisted of non-drug users with fungal infections
  Direct Examination: It was an observational study and subjects received their routine treatment.
Period: Overall Study
Arm/Group | Drug Users | Non-drug Users
Started | 718 | 718
Completed | 73 | 62
Not Completed | 645 | 656

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug Users | Non-drug Users | Total
Number analyzed (Participants) | 718 | 718 | 1436
Age, Continuous [Mean (Full Range); unit: years] | 38.3 [9 to 90] | 36.8 [11 to 86] | 37.55 [9 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 137 | 253
  Male | 602 | 581 | 1183
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 718 | 718 | 1436

OUTCOME MEASURES:

1. Primary Outcome: The Prevalence of Superficial and Cutaneous Fungal Infections Among Drug and Non-Drug Users
Time Frame: up to two months
Measure: Number; unit: participants
Arm/Group | Drug Users | Non-drug Users
Number analyzed (Participants) | 718 | 718
participants | 73 | 62

ADVERSE EVENTS:
Description: Serious and Other Adverse Events were not collected
Arm/Group | Drug Users | Non-drug Users
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes